CLINICAL TRIAL: NCT05960045
Title: Testing Tolerance in Cow Milk Protein Allergy Patients: Milk Ladder or Direct Milk Administration?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: MS 476/2021
Record Dates: First submitted 2022-09-10; First posted 2023-07-25 (Actual); Last update posted 2025-05-07 (Actual); Status verified 2025-04

CONDITIONS: Cow Milk Allergy; Tolerance
MeSH Terms: conditions — Milk Hypersensitivity

STUDY DESIGN:
Intervention Model Description: 2 groups
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Patients receiving direct milk antigen (Group A) (Active Comparator): Patients with cow milk protein allergy after 6 month of elimination diet will receive direct milk antigen and will be followed up for 2 months for the development of any symptoms of milk intolerance
  Interventions: Dietary Supplement: Direct Milk antigen reintroduction
- Patients subjected to gradual reintroduction of milk through a milk ladder (Group B) (Active Comparator): Patient with cow milk protein allergy after 6 month of elimination diet will be offered indirect milk antigen through a ladder starting by baked milk products and will be followed up for also for 2 months to detect any symptoms of intolerance.
  Interventions: Dietary Supplement: Milk ladder

INTERVENTIONS:
Dietary Supplement: Direct Milk antigen reintroduction — Direct milk antigen re-introduction milk according to ESPGHAN guidelines
  Arms: Patients receiving direct milk antigen (Group A)
Dietary Supplement: Milk ladder — B: Milk ladder according to the iMAP guideline which are 6 weeks of gradual reintroduction starting with baked milk not direct antigen
  Arms: Patients subjected to gradual reintroduction of milk through a milk ladder (Group B)

SUMMARY:
Majority of children outgrow their allergies, however there are two different methods to re-introduce milk products in the infant diet either direct milk intake in escalating doses or milk ladder, starting with baked milk products instead of pure milk.

This study aims to compare rate of tolerance after milk reintroduction among patient with cow milk protein allergy (CMPA) diagnosed by elimination re-challenge test after six months of elimination diet by milk ladder versus direct milk intake.

DETAILED DESCRIPTION:
CMPA is an immunological response to one or more milk proteins. CMPA may be IgE mediated or Non-IgE mediated. It is one of the most frequent causes of food allergies in young children with an estimated prevalence between 1.9% and 4.9% in the first year of life.

CMPA has a good prognosis and cow milk is reintroduced in child diet. Natural history of CMPA shows heterogeneity and it is closely related to the clinical phenotype by which it was presented.

The timing and evaluation of developing tolerance is determined by clinical response to milk introduction.

When diagnosis of CMPA is confirmed, fresh pasteurized cow's milk can be used above 12 months of age in oral food challenge procedure, the starting dose should be lower than a dose that can induce a reaction and then increased step wise to 100ml, in children with mild to moderate reactions doses of 1ml, 3ml, 10ml, 30ml, and 100ml may be given at 30 minutes' intervals.

The milk ladder is an evidence-based plan to re-introduce milk products gradually and in stages for infants and children with mild to moderate cow's milk allergy, starting with food that contain only small amount of well-cooked milk and progressing towards uncooked dairy products and fresh milk. It's only started once child has been on a milk free diet for at least 6 months and they are completely well with no active eczema or gastro-intestinal symptoms.

Addition of baked- milk to the diet appears to accelerate the development of unheated-milk tolerance compared to strict avoidance, also its consumption is considered a form of immunotherapy with favorable safety, higher convenience, lower cost and less intensity when compared to oral immunotherapy. It's suggested to enhance the quality of life by removing unnecessary dietary restrictions and change the natural evaluation of milk allergy by promoting the development of tolerance to regular cow's milk.

ELIGIBILITY:
Inclusion Criteria:

1. Patients age between 9 months old till 3 years old.
2. Patients with symptoms that suggest mild to moderate non IgE mediated Cow Milk Allergy
3. Patients on strict elimination diet for at least six months duration

Exclusion Criteria:

Patient with:

* Chronic gastrointestinal disease (malabsorption, irritable bowel syndrome).
* Multiple food allergy and/or history of anaphylaxis.
* Ongoing eczema or severe gastrointestinal symptoms.

Ages: 9 Months to 3 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 116 (Actual)
Dates: Start 2024-07-01 (Actual); Primary Completion 2025-04-15 (Actual); Study Completion 2025-04-28 (Actual)

PRIMARY OUTCOMES:
Compare the frequency of tolerance to milk between the two groups | intervention will be made six months of elimination diet, and follow up of 2 months later
  Questionnaire done to assess occurrence of following symptoms Vomiting, Hematemesis, Diarrhea (using BRISTOL scale), Constipation, Eczema, Skin rash, Perianal inflammation, weight loss in kilograms or failure to gain weight in kilograms, (Colic, Straining and marked Abdominal distension), and recurrent respiratory symptoms within two months of following up after milk reintroduction. If any of the previous items is present, then the patient is considered intolerant to milk. All items should be answered by (no) in order to consider the patient tolerant to milk

SECONDARY OUTCOMES:
Recording of overall percentage of milk tolerance after 6 months elimination diet | intervention will be made six months of elimination diet, and follow up of 2 months later
  the same questionnaire used to assess tolerance to milk products. Also all answers should be answered by No, otherwise patient would still be considered intolerant.

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Saber, Study Director — AinShams University; Yasmine El-Gendy, Study Director — AinShams university; Yosra Awad, Study Director — Ain Shams University; Nesreen Hammad, Study Director — Ain Shams University; Mostafa EL-Hodhod, Principal Investigator — Ain Shams University
Locations (1):
- Ain Shams University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bahna SL. Cow's milk allergy versus cow milk intolerance. Ann Allergy Asthma Immunol. 2002 Dec;89(6 Suppl 1):56-60. doi: 10.1016/s1081-1206(10)62124-2. PMID 12487206
- [Background] NIAID-Sponsored Expert Panel; Boyce JA, Assa'ad A, Burks AW, Jones SM, Sampson HA, Wood RA, Plaut M, Cooper SF, Fenton MJ, Arshad SH, Bahna SL, Beck LA, Byrd-Bredbenner C, Camargo CA Jr, Eichenfield L, Furuta GT, Hanifin JM, Jones C, Kraft M, Levy BD, Lieberman P, Luccioli S, McCall KM, Schneider LC, Simon RA, Simons FE, Teach SJ, Yawn BP, Schwaninger JM. Guidelines for the diagnosis and management of food allergy in the United States: report of the NIAID-sponsored expert panel. J Allergy Clin Immunol. 2010 Dec;126(6 Suppl):S1-58. doi: 10.1016/j.jaci.2010.10.007. PMID 21134576
- [Background] Esmaeilzadeh H, Alyasin S, Haghighat M, Nabavizadeh H, Esmaeilzadeh E, Mosavat F. The effect of baked milk on accelerating unheated cow's milk tolerance: A control randomized clinical trial. Pediatr Allergy Immunol. 2018 Nov;29(7):747-753. doi: 10.1111/pai.12958. Epub 2018 Sep 12. PMID 30027590
- [Background] Fiocchi A, Schunemann HJ, Brozek J, Restani P, Beyer K, Troncone R, Martelli A, Terracciano L, Bahna SL, Rance F, Ebisawa M, Heine RG, Assa'ad A, Sampson H, Verduci E, Bouygue GR, Baena-Cagnani C, Canonica W, Lockey RF. Diagnosis and Rationale for Action Against Cow's Milk Allergy (DRACMA): a summary report. J Allergy Clin Immunol. 2010 Dec;126(6):1119-28.e12. doi: 10.1016/j.jaci.2010.10.011. PMID 21134569
- [Background] Kim JS, Nowak-Wegrzyn A, Sicherer SH, Noone S, Moshier EL, Sampson HA. Dietary baked milk accelerates the resolution of cow's milk allergy in children. J Allergy Clin Immunol. 2011 Jul;128(1):125-131.e2. doi: 10.1016/j.jaci.2011.04.036. Epub 2011 May 23. PMID 21601913
- [Background] Koletzko S, Niggemann B, Arato A, Dias JA, Heuschkel R, Husby S, Mearin ML, Papadopoulou A, Ruemmele FM, Staiano A, Schappi MG, Vandenplas Y; European Society of Pediatric Gastroenterology, Hepatology, and Nutrition. Diagnostic approach and management of cow's-milk protein allergy in infants and children: ESPGHAN GI Committee practical guidelines. J Pediatr Gastroenterol Nutr. 2012 Aug;55(2):221-9. doi: 10.1097/MPG.0b013e31825c9482. PMID 22569527
- [Background] Lambert R, Grimshaw KEC, Ellis B, Jaitly J, Roberts G. Evidence that eating baked egg or milk influences egg or milk allergy resolution: a systematic review. Clin Exp Allergy. 2017 Jun;47(6):829-837. doi: 10.1111/cea.12940. Epub 2017 May 17. PMID 28516451
- [Background] Longo G, Barbi E, Berti I, Meneghetti R, Pittalis A, Ronfani L, Ventura A. Specific oral tolerance induction in children with very severe cow's milk-induced reactions. J Allergy Clin Immunol. 2008 Feb;121(2):343-7. doi: 10.1016/j.jaci.2007.10.029. Epub 2007 Dec 26. PMID 18158176
- [Background] Luyt D, Ball H, Makwana N, Green MR, Bravin K, Nasser SM, Clark AT; Standards of Care Committee (SOCC) of the British Society for Allergy and Clinical Immunology (BSACI). BSACI guideline for the diagnosis and management of cow's milk allergy. Clin Exp Allergy. 2014;44(5):642-72. doi: 10.1111/cea.12302. PMID 24588904
- [Background] Nicolaou N, Tsabouri S, Priftis KN. Reintroduction of cow's milk in milk-allergic children. Endocr Metab Immune Disord Drug Targets. 2014 Mar;14(1):54-62. doi: 10.2174/1871530314666140121150228. PMID 24450449
- [Background] Niggemann B, Beyer K. Diagnosis of food allergy in children: toward a standardization of food challenge. J Pediatr Gastroenterol Nutr. 2007 Oct;45(4):399-404. doi: 10.1097/MPG.0b013e318054b0c3. PMID 18030203
- [Background] Upton J, Nowak-Wegrzyn A. The Impact of Baked Egg and Baked Milk Diets on IgE- and Non-IgE-Mediated Allergy. Clin Rev Allergy Immunol. 2018 Oct;55(2):118-138. doi: 10.1007/s12016-018-8669-0. PMID 29516263
- [Background] Vandenplas Y, Koletzko S, Isolauri E, Hill D, Oranje AP, Brueton M, Staiano A, Dupont C. Guidelines for the diagnosis and management of cow's milk protein allergy in infants. Arch Dis Child. 2007 Oct;92(10):902-8. doi: 10.1136/adc.2006.110999. PMID 17895338
- [Background] Venter C, Brown T, Meyer R, Walsh J, Shah N, Nowak-Wegrzyn A, Chen TX, Fleischer DM, Heine RG, Levin M, Vieira MC, Fox AT. Better recognition, diagnosis and management of non-IgE-mediated cow's milk allergy in infancy: iMAP-an international interpretation of the MAP (Milk Allergy in Primary Care) guideline. Clin Transl Allergy. 2017 Aug 23;7:26. doi: 10.1186/s13601-017-0162-y. eCollection 2017. PMID 28852472
- [Background] Yang M, Tan M, Wu J, Chen Z, Long X, Zeng Y, Cai H, Zhang Y, Geng L, Xiao Y, Ke H, Liu Y, Rong L, Fu S, Wang H, Wang Y, Li X, Chen P, Li K, Xie J, Chen H, Li H, Wang H, Li DY, Gong S. Prevalence, Characteristics, and Outcome of Cow's Milk Protein Allergy in Chinese Infants: A Population-Based Survey. JPEN J Parenter Enteral Nutr. 2019 Aug;43(6):803-808. doi: 10.1002/jpen.1472. Epub 2018 Nov 19. PMID 30452099